CLINICAL TRIAL: NCT01700205
Title: Impact of Diet Composition on Energy Balance and Satiety During Infancy
Brief Title: Effect of Infant Formula on Energy Balance
Acronym: GRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: University of Delaware (Other); Children's Hospital of Philadelphia (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Julie A. Mennella, PhD, Member, Monell Chemical Senses Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HD072307
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Development
Keywords: Formula Feeding; Mother; Moms; Infants; Babies; Baby; growth; energy balance

STUDY DESIGN:
Intervention Model Description: Between- and within-subject longitudinal trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type of Formula: CMF (Active Comparator): Infants are randomized to feed standard cow milk formula during first year of life
  Interventions: Other: Type of Formula
- Type of Formula: EHF (Experimental): Infants are randomized to feed extensively hydrolyzed infant formula during first year of life
  Interventions: Other: Type of Formula

INTERVENTIONS:
Other: Type of Formula — infant formula
  Other Names: cow milk formula (CMF); protein hydrolysate formula (EHF)

SUMMARY:
The overarching goal of the research we propose here is to conduct a randomized clinical trial to specify the physiologic and behavioral mechanisms by which infant-formula composition affects all aspects of energy balance and growth during the first years of life.

DETAILED DESCRIPTION:
This is a randomized clinical trial of infants whose parents decided to formula feed them; mother-infant dyads will be randomized when infant is 2 weeks of age to one of 2 groups. The groups will differ in the composition of the formula fed to the infant during the first year of life.

ELIGIBILITY:
Inclusion Criteria

1. A healthy, term (≥37 and ≤42 week gestation at birth), singleton infant.
2. Birth weight between 2500 - 4500 grams.
3. At the time of enrollment, infant must be ≤14 days old (Date of birth=day 0).
4. Mother must be 18 years or older.
5. Infant must be consuming a standard cow's milk protein infant formula and have been receiving a standard cow's milk protein infant formula for at least the past 2 days prior to enrollment.

Exclusion Criteria

1. Mother had gestational diabetes during pregnancy
2. Infant has condition requiring infant feedings other than feeding cow milk formula from a bottle.
3. Infant has major congenital malformations (i.e. cleft palate, hemangiomas, extremity malformation).
4. Infant has suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus).
5. Infant has evidence of significant cardiac, respiratory, endocrinologic, hematologic, gastrointestinal, or other systemic diseases. For example, infant must not be receiving insulin or growth hormone.
6. Dyad be the relative (son, daughter, niece, nephew, cousin, aunt, uncle, sibling) of ancillary personnel connected with the study.

Ages: 1 Week to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center; Jillian Trabulsi, PhD, Principal Investigator — University of Delaware
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Energy balance measures at 0.75, 3.5 and 12.5 months of age

REFERENCES:
- [Background] Mennella JA, Ventura AK, Beauchamp GK. Differential growth patterns among healthy infants fed protein hydrolysate or cow-milk formulas. Pediatrics. 2011 Jan;127(1):110-8. doi: 10.1542/peds.2010-1675. Epub 2010 Dec 27. PMID 21187303
- [Background] Mennella JA, Beauchamp GK. Developmental changes in the acceptance of protein hydrolysate formula. J Dev Behav Pediatr. 1996 Dec;17(6):386-91. doi: 10.1097/00004703-199612000-00003. PMID 8960567
- [Background] Mennella JA, Lukasewycz LD, Castor SM, Beauchamp GK. The timing and duration of a sensitive period in human flavor learning: a randomized trial. Am J Clin Nutr. 2011 May;93(5):1019-24. doi: 10.3945/ajcn.110.003541. Epub 2011 Feb 10. PMID 21310829
- [Result] Mennella JA, Inamdar L, Pressman N, Schall JI, Papas MA, Schoeller D, Stallings VA, Trabulsi JC. Type of infant formula increases early weight gain and impacts energy balance: a randomized controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):1015-1025. doi: 10.1093/ajcn/nqy188. PMID 30295700
- [Result] Mennella JA, Papas MA, Reiter AR, Stallings VA, Trabulsi JC. Early rapid weight gain among formula-fed infants: Impact of formula type and maternal feeding styles. Pediatr Obes. 2019 Jun;14(6):e12503. doi: 10.1111/ijpo.12503. Epub 2019 Jan 10. PMID 30629845
- [Derived] Decker JE, Mennella JA, Brewer BC, Robson SM, Millen AE, Delahanty MT, Smethers AD, Trabulsi JC. Association Between Diet Patterns of Human Infants and Growth Differs Across Randomized Formula Groups in the First 18.5 Months. J Nutr. 2025 Dec;155(12):4390-4400. doi: 10.1016/j.tjnut.2025.10.007. Epub 2025 Oct 11. PMID 41082983
- [Derived] Mennella JA, Smethers AD, Delahanty MT, Stallings VA, Trabulsi JC. Glutamic Acid Intake by Formula-Fed Infants: Are Acceptable Daily Intakes Feasible? Res Sq [Preprint]. 2023 May 17:rs.3.rs-2907953. doi: 10.21203/rs.3.rs-2907953/v1. PMID 37292800
- [Derived] Mennella JA, Reiter A, Brewer B, Pohlig RT, Stallings VA, Trabulsi JC. Early Weight Gain Forecasts Accelerated Eruption of Deciduous Teeth and Later Overweight Status during the First Year. J Pediatr. 2020 Oct;225:174-181.e2. doi: 10.1016/j.jpeds.2020.06.019. Epub 2020 Jun 15. PMID 32553836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2012 to 2015, newly parturient women whose decision not to lactate was firmly established were recruited through ads in regional newspapers, websites and hospitals in the greater Philadelphia area.
Groups:
- Type of Formula: CMF: infant is randomized to feed standard cow milk formula during first year of life
  Type of Formula: infant formula
- Type of Formula: EHF: infant is randomized to feed extensively hydrolyzed infant formula during first year of life
  Type of Formula: infant formula
Period: Overall Study
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Started | 59 (Mother-Infant Dyads) | 54 (Mother-Infant Dyads)
Completed | 44 (Mother-Infant Dyads) | 39 (Mother-Infant Dyads)
Not Completed | 15 | 15
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Type of Formula: CMF: infant is randomized to feed standard cow milk infant formula [CMF] during first year of life
  Type of Formula: infant formula
- Type of Formula: EHF: infant is randomized to feed extensively hydrolyzed protein infant formula [EHF] first year of life
  Type of Formula: infant formula
- Total: Total of all reporting groups
Arm/Group | Type of Formula: CMF | Type of Formula: EHF | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Continuous [Mean (Standard Deviation); unit: Months] | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 31 | 25 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 54 | 46 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 35 | 70
  White | 17 | 8 | 25
  More than one race | 7 | 11 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 54 | 113
TAS2R38 genotype, A49P allele; infants [Count of Participants; unit: Participants]
  AA, homozygous recessive | 19 | 15 | 34
  AP, heterozygous | 27 | 25 | 52
  PP, homozygous dominant | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Growth, Weight for Length (WLZ) Z Scores
Description: At each visit, infants were weighed and measured to monitor normal growth. These anthropometric data were converted to weight-for-length (WLZ) Zscores using World Health Organization (WHO) growth standards. The Z-score expresses the anthropometric value as a number of standard deviations or Z-scores below or above the reference mean value. Normal range for Z score is -2.0 (minimum) to 2.0 (maximum).
Time Frame: 0.5 to 12.5 months with followup visit at 18.5 mos
Population: We conducted an intention-to-treat (ITT) analyses on 113 infants regardless of study withdrawal.
Measure: Mean (Standard Error); unit: Z score
Groups:
- Type of Formula: CMF: Infant is randomized to be fed standard cow milk formula during first year of life
  Type of Formula: CMF
- Type of Formula: EHF: Infant is randomized to be fed extensively protein hydrolyzed infant formula during first year of life
  Type of Formula: EHF
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
Z score
  Weight for Length Z, 0.5 mos | -0.26 (0.13) | -0.12 (0.13)
  Weight for Length Z, 0.75 mos | -0.12 (0.13) | 0.13 (0.13)
  Weight for Length Z, 1.5 mos: number analyzed (Participants) | 57 | 52
  Weight for Length Z, 1.5 mos | 0.24 (0.13) | -0.17 (0.13)
  Weight for Length Z, 2.5 mos: number analyzed (Participants) | 55 | 52
  Weight for Length Z, 2.5 mos | 0.24 (0.13) | -0.17 (0.13)
  Weight for Length Z, 3.5 mos: number analyzed (Participants) | 53 | 48
  Weight for Length Z, 3.5 mos | 0.22 (0.13) | -0.38 (0.14)
  Weight for Length Z, 4.5 mos: number analyzed (Participants) | 48 | 44
  Weight for Length Z, 4.5 mos | 0.39 (0.13) | -0.24 (0.14)
  Weight for Length Z, 5.5 mos: number analyzed (Participants) | 46 | 44
  Weight for Length Z, 5.5 mos | 0.42 (0.14) | -0.36 (0.14)
  Weight for Length Z, 6.5 mos: number analyzed (Participants) | 46 | 44
  Weight for Length Z, 6.5 mos | 0.52 (0.14) | 0.18 (0.14)
  Weight for Length Z, 7.5 mos: number analyzed (Participants) | 46 | 43
  Weight for Length Z, 7.5 mos | 0.59 (0.14) | 0.20 (0.14)
  Weight for Length Z, 8.5 mos: number analyzed (Participants) | 46 | 43
  Weight for Length Z, 8.5 mos | 0.76 (0.14) | 0.29 (0.14)
  Weight for Length Z, 9.5 mos: number analyzed (Participants) | 46 | 42
  Weight for Length Z, 9.5 mos | 0.71 (0.14) | 0.40 (0.14)
  Weight for Length Z, 10.5 mos: number analyzed (Participants) | 46 | 40
  Weight for Length Z, 10.5 mos | 0.76 (0.14) | 0.46 (0.14)
  Weight for Length Z, 11.5 mos: number analyzed (Participants) | 45 | 40
  Weight for Length Z, 11.5 mos | 0.72 (0.14) | 0.51 (0.14)
  Weight for Length Z, 12.5 mos: number analyzed (Participants) | 44 | 39
  Weight for Length Z, 12.5 mos | 0.70 (0.14) | 0.52 (0.14)
  Weight for Length Z, 18.5 mos: number analyzed (Participants) | 40 | 38
  Weight for Length Z, 18.5 mos | 0.80 (0.14) | 0.68 (0.15)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Test type: Other — A priori power analyses determined that a sample size of 94 is required to detect a difference of 0.67 with 90% power and a 5% type 1 error rate. We conducted an intention-to-treat (ITT) analyses on the 113 infants using separate generalized estimating equations that included treatment group (CMF, EHF), time (infant age), and group × time interaction for each type of Z score (0.5-12.5 mos); p < 0.05, Generalized Estimating Equation; GEE analysis conducted with group (CMF, EHF), time (infant age, 0.5-12.5 months) and their interaction; Slope = -0.018, 95% CI 2-sided [-0.0363 to -0.0002]

2. Primary Outcome: Growth, Weight for Age (WAZ) Z Score
Description: At each visit, infants were weighed to monitor normal growth. These anthropometric data were converted to Weight for age Z (WAZ) Z scores using World Health Organization (WHO) growth standards. The Z-score expresses the anthropometric value as a number of standard deviations or Z-scores below or above the reference mean value. Normal range for Z score is -2.0 (minimum) to 2.0 (maximum).
Time Frame: 0.5 to 12.5 months with followup visit at 18.5 mos
Population: We conducted an intention-to-treat (ITT) analyses on 113 infants regardless of study withdrawal.
Measure: Mean (Standard Error); unit: Z score
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
Z score
  Weight for Age Z score, 0.5 mos | -0.36 (0.12) | -0.25 (0.13)
  Weight for Age Z score, 0.75 mos | -0.41 (0.12) | -0.28 (0.13)
  Weight for Age Z score, 1.5 mos: number analyzed (Participants) | 57 | 52
  Weight for Age Z score, 1.5 mos | -0.38 (0.12) | -0.61 (0.13)
  Weight for Age Z score, 2.5 mos: number analyzed (Participants) | 55 | 53
  Weight for Age Z score, 2.5 mos | -0.34 (0.12) | -0.66 (0.13)
  Weight for Age Z score, 3.5 mos: number analyzed (Participants) | 53 | 49
  Weight for Age Z score, 3.5 mos | -0.14 (0.12) | 0.64 (0.13)
  Weight for Age Z score, 4.5 mos: number analyzed (Participants) | 48 | 44
  Weight for Age Z score, 4.5 mos | 0.07 (0.13) | -0.37 (0.13)
  Weight for Age Z score, 5.5 mos: number analyzed (Participants) | 46 | 44
  Weight for Age Z score, 5.5 mos | 0.18 (0.13) | -0.20 (0.13)
  Weight for Age Z score, 6.5 mos: number analyzed (Participants) | 48 | 44
  Weight for Age Z score, 6.5 mos | 0.29 (0.13) | -0.03 (0.13)
  Weight for Age Z score, 7.5 mos: number analyzed (Participants) | 46 | 43
  Weight for Age Z score, 7.5 mos | 0.38 (0.13) | 0.02 (0.13)
  Weight for Age Z score, 8.5 mos: number analyzed (Participants) | 46 | 43
  Weight for Age Z score, 8.5 mos | 0.50 (0.13) | 0.08 (0.13)
  Weight for Age Z score, 9.5 mos: number analyzed (Participants) | 47 | 42
  Weight for Age Z score, 9.5 mos | 0.51 (0.13) | 0.16 (0.13)
  Weight for Age Z score, 10.5 mos: number analyzed (Participants) | 47 | 40
  Weight for Age Z score, 10.5 mos | 0.54 (0.13) | 0.20 (0.13)
  Weight for Age Z score, 11.5 mos: number analyzed (Participants) | 45 | 40
  Weight for Age Z score, 11.5 mos | 0.52 (0.13) | 0.28 (0.13)
  Weight for Age Z score, 12.5 mos: number analyzed (Participants) | 44 | 39
  Weight for Age Z score, 12.5 mos | 0.52 (0.13) | 0.32 (0.13)
  Weight for Age Z score, 18.5 mos: number analyzed (Participants) | 40 | 38
  Weight for Age Z score, 18.5 mos | 0.56 (0.14) | 0.40 (0.15)
  Length for Age Z score, 18.5 mos: number analyzed (Participants) | 40 | 38
  Length for Age Z score, 18.5 mos | -0.07 (0.14) | -0.22 (0.16)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Test type: Other — A priori power analyses determined that a sample size of 94 is required to detect a difference of 0.67 with 90% power and a 5% type 1 error rate. We conducted an intention-to-treat (ITT) analyses on the 113 infants using separate generalized estimating equations that included treatment group (CMF, EHF), time (infant age), and group × time interaction for each type of Z score (0.5-12.5 mos). We provide below the parameter estimates for WLZ scores only; p = 0.001, Generalized Estimating Equations; GEE analysis conducted on each type of Z score separately with group (CMF, EHF), time (infant age; 0.5-12.5 months) and their interaction; Slope = -0.023, 95% CI 2-sided [-0.0362 to -0.0093]

3. Primary Outcome: Growth: Length for Age (LAZ) Z Scores
Description: At each visit, infants were measured to monitor normal growth. These anthropometric data were converted to Length for age Z (LAZ) Z scores using World Health Organization (WHO) growth standards. The Z-score expresses the anthropometric value as a number of standard deviations or Z-scores below or above the reference mean value. Normal range for Z score is -2.0 (minimum) to 2.0 (maximum).
Time Frame: 0.5 to 12.5 months with followup visit at 18.5 mos
Population: We conducted an intention-to-treat (ITT) analyses on 113 infants regardless of study withdrawal.
Measure: Mean (Standard Error); unit: Z score
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
Z score
  Length for Age Z score, 0.5 mos | -0.49 (0.14) | -0.46 (0.14)
  Length for Age Z score, 0.75 mos | -0.56 (0.14) | 0.59 (0.14)
  Length for Age Z score, 1.5 mos: number analyzed (Participants) | 57 | 52
  Length for Age Z score, 1.5 mos | -0.55 (0.14) | -0.48 (0.14)
  Length for Age Z score, 2.5 mos: number analyzed (Participants) | 55 | 52
  Length for Age Z score, 2.5 mos | -0.57 (0.14) | -0.62 (0.14)
  Length for Age Z score, 3.5mos: number analyzed (Participants) | 53 | 48
  Length for Age Z score, 3.5mos | -0.36 (0.14) | -0.43 (0.15)
  Length for Age Z score, 4.5 mos: number analyzed (Participants) | 48 | 44
  Length for Age Z score, 4.5 mos | -0.26 (0.14) | -0.21 (0.15)
  Length for Age Z score, 5.5 mos: number analyzed (Participants) | 46 | 44
  Length for Age Z score, 5.5 mos | -0.13 (0.14) | -0.17 (0.15)
  Length for Age Z score, 6.5 mos: number analyzed (Participants) | 46 | 44
  Length for Age Z score, 6.5 mos | -0.05 (0.14) | -0.17 (0.15)
  Length for Age Z score, 7.5 mos: number analyzed (Participants) | 46 | 43
  Length for Age Z score, 7.5 mos | 0.01 (0.14) | -0.11 (0.15)
  Length for Age Z score, 8.5 mos: number analyzed (Participants) | 46 | 43
  Length for Age Z score, 8.5 mos | -0.02 (0.14) | -0.16 (0.15)
  Length for Age Z score, 9.5 mos: number analyzed (Participants) | 46 | 42
  Length for Age Z score, 9.5 mos | 0.01 (0.14) | -0.19 (0.15)
  Length for Age Z score, 10.5 mos: number analyzed (Participants) | 46 | 40
  Length for Age Z score, 10.5 mos | 0.01 (0.14) | -0.21 (0.15)
  Length for Age Z score, 11.5 mos: number analyzed (Participants) | 45 | 40
  Length for Age Z score, 11.5 mos | 0.00 (0.14) | -0.18 (0.15)
  Length for Age Z score, 12.5 mos: number analyzed (Participants) | 44 | 39
  Length for Age Z score, 12.5 mos | 0.03 (0.14) | -0.13 (0.15)
  Length for Age Z score, 18.5 mos: number analyzed (Participants) | 40 | 38
  Length for Age Z score, 18.5 mos | -0.07 (0.14) | -0.22 (0.16)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.32, Generalized Estimating Equation; GEE analysis conducted with group (CMF, EHF), time (infant age, 0.5-12.5 months) and their interaction; Slope = -0.02, 95% CI 2-sided [-0.058 to 0.019]

4. Primary Outcome: Energy Balance: Energy Intake From Infant Formula and Other Sources
Description: Energy intake (kcal/day) of infant formula and other sources was determined by three-day weighed bottle intake and records of the infants' intake of any liquid or food other than formula during the three days
Time Frame: 0.75, 3.5, 12.5 mos
Population: Intent-to-treat analysis (N=113).
Measure: Mean (Standard Error); unit: kcal per day
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
kcal per day
  Energy Intake from Formula, 0.75 months: number analyzed (Participants) | 52 | 46
  Energy Intake from Formula, 0.75 months | 466 (14) | 383 (15)
  Energy Intake from Other Sources, 0.75 months: number analyzed (Participants) | 52 | 46
  Energy Intake from Other Sources, 0.75 months | 0 (0) | 0 (0)
  Energy Intake from Formula, 3.5 mos: number analyzed (Participants) | 36 | 32
  Energy Intake from Formula, 3.5 mos | 628 (21) | 596 (21)
  Energy Intake from Other Sources, 3.5 mos: number analyzed (Participants) | 36 | 32
  Energy Intake from Other Sources, 3.5 mos | 11 (5) | 10 (6)
  Energy Intake from Formula, 12.5 mos: number analyzed (Participants) | 36 | 30
  Energy Intake from Formula, 12.5 mos | 425 (50) | 284 (56)
  Energy Intake from Other Sources, 12.5 mos: number analyzed (Participants) | 36 | 30
  Energy Intake from Other Sources, 12.5 mos | 712 (51) | 863 (57)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; ANOVAs were conducted with group (CMF, EHF) as the between-subjects factor; Test type: Other — ANOVA with group (CMF, EHF) as between-subjects factor were conducted on intent-to-treat sample; p < 0.05, Repeated Measures ANOVA; We conducted a ANOVA with group (CMF, EHF) as between-subject factor

5. Primary Outcome: Energy Balance: Sleeping Energy Expenditure (SEE)
Description: Postprandial SEE (kcal/day), a proxy for resting energy expenditure in infant, was measured for a minimum of 30 min by open-circuit, indirect calorimetry using a metabolic cart with canopy hood, in a quiet, thermal-neutral room.
Time Frame: 0.75, 3.5, 12.5 mos
Population: Intent-to-treat analysis (N=113).
Measure: Mean (Standard Error); unit: kcal per day
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
kcal per day
  Sleeping Energy Expenditure (0.75 months): number analyzed (Participants) | 54 | 48
  Sleeping Energy Expenditure (0.75 months) | 206 (6) | 201 (6)
  Sleeping Energy Expenditure, 3.5 months: number analyzed (Participants) | 47 | 42
  Sleeping Energy Expenditure, 3.5 months | 329 (8) | 321 (8)
  Sleeping Energy Expenditure, 12.5 months: number analyzed (Participants) | 36 | 35
  Sleeping Energy Expenditure, 12.5 months | 507 (11) | 509 (11)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor; Test type: Other — ANOVA was conducted with group (CMF, EHF) as between-subjects factor on the intent-to-treat sample; p = 0.72, Repeated Measure ANOVA; ANOVA was conducted with group (CMF, EHF) as between-subjects factor on the intent-to-treat sample

6. Primary Outcome: Energy Balance: Total Energy Expenditure (TEE)
Description: TEE (kcal/day) was measured over 7 days at each of the three time points (0.75, 3.5 and12.5 mos) using the doubly labeled water method
Time Frame: 0.75, 3.5, 12.5 mos
Population: Intent-to-treat analysis (N=113).
Measure: Mean (Standard Error); unit: kcal per day
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
kcal per day
  Total energy expenditure, 0.75 months: number analyzed (Participants) | 55 | 39
  Total energy expenditure, 0.75 months | 283 (18) | 243 (19)
  Total energy expenditure, 3.5 months: number analyzed (Participants) | 45 | 39
  Total energy expenditure, 3.5 months | 488 (24) | 444 (26)
  Total energy expenditure, 12.5 months: number analyzed (Participants) | 29 | 29
  Total energy expenditure, 12.5 months | 859 (42) | 858 (45)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample; Test type: Other — Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample; p = 0.72, Repeated Measure ANOVA; Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample

7. Primary Outcome: Energy Balance: Energy Loss in Stools
Description: Stool EL (kcal/day) was determined from 3-day stool collection by bomb calorimetry at each timepoint
Time Frame: 0.75, 3.5, 12.5 mos
Population: Intent-to-treat analysis (N=113).
Measure: Mean (Standard Error); unit: kcal per day
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
kcal per day
  Energy Loss in Stools, 0.75 months: number analyzed (Participants) | 56 | 44
  Energy Loss in Stools, 0.75 months | 22.3 (3.9) | 34.9 (4.1)
  Energy Loss in Stools, 3.5 months: number analyzed (Participants) | 46 | 42
  Energy Loss in Stools, 3.5 months | 20.7 (1.8) | 17.0 (1.9)
  Energy Loss in Stools, 12.5 months: number analyzed (Participants) | 36 | 36
  Energy Loss in Stools, 12.5 months | 27.1 (3.2) | 33.8 (3.4)
Statistical Analysis 1: Comparison: Type of Formula: CMF vs Type of Formula: EHF; Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample; Test type: Other — Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample; p = 0.02, Repeated Measure ANOVA; Repeated Measures ANOVA conducted with group (CMF, EHF) as between-subjects factor on intent-to-treat sample

8. Secondary Outcome: Feeding Behaviors, Maternal Perceptions
Description: Maternal perception of infant feeding behavior, using standardized questionnaires (Infant feeding style questionnaire; IFSQ); values ranged from 1 to 5; higher scores reflect more of that feeding style. Only baseline data reported herein.
Time Frame: 0.5 months
Population: Some mothers responded N/A on questions related to restrictive feeding styles and thus score for this subscale could not be computed.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
Number analyzed (Participants) | 59 | 54
Units on a scale
  Laissez-Faire Feeding Style, 0.5 mos | 3.1 (0.1) | 3.0 (0.1)
  Restrictive Feeding Style, 0.5 mos: number analyzed (Participants) | 52 | 46
  Restrictive Feeding Style, 0.5 mos | 2.8 (0.1) | 2.6 (0.2)
  Pressure to Eat Feeding Style, 0.5 mos | 2.2 (0.1) | 2.4 (0.1)
  Responsive Feeding Styly, 0.5 mos | 4.1 (0.1) | 4.0 (0.1)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Type of Formula: CMF | Type of Formula: EHF
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/54
Other Adverse Events (participants affected / at risk) | 0/59 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No